CLINICAL TRIAL: NCT00735618
Title: Pilot Study on the Effects of a Brief Relaxation Program on Heart Rate Variability in Cancer Patients
Brief Title: Relaxation and Heart Rate Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0028
Record Dates: First submitted 2008-08-12; First posted 2008-08-15 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-11

CONDITIONS: Cancer
Keywords: Advanced Cancer; Cancer Patients; Relaxation Therapy; Relaxation and Heart Rate Variability; Guided Relaxation; HRV; Stress, Anxiety, and Panic Disorder
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Panic Disorder | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Guided Relaxation (Experimental): Heart rate variability (HRV) high frequency (HF) spectral analysis, before and after a 15 minute, one-time, guided relaxation program
  Interventions: Other: Guided Relaxation

INTERVENTIONS:
Other: Guided Relaxation — Following 5 minute questionnaire, 15 minute rest and 5 minute heart rhythm recording, 15 minute relaxation program (listening via headphone to audio recording) to be completed by second heart rhythm recording and same questionnaire. Entire procedure 45-60 minutes.
  Other Names: Relaxation Therapy; Guided Relaxation Program

SUMMARY:
Primary:

* To characterize the physiologic changes of the autonomic nervous system, demonstrated by heart rate variability (HRV) high frequency (HF) spectral analysis, before and after a 15 minute, one-time, guided relaxation program for cancer patients.

Secondary:

* To assess whether change of HRV correlates with subjective feeling for anxiety, based on visual analog scale scores.

DETAILED DESCRIPTION:
Rhythm changes in your heart rate are part of the "autonomic" nervous system. This is the part of your nervous system that controls the body functions that you do not have to think about. Researchers want to find out if a "guided relaxation" session will make your heart rate more variable, with more rhythm changes.

If you are found to be eligible to take part in this study, you will first answer a brief questionnaire that will measure several symptoms, such as pain and anxiety (worry). This questionnaire will take less than 5 minutes. You will also be asked questions about your alcohol and smoking history, and if you have ever used relaxation or meditation techniques in the past. This will also take less than 5 minutes.

You will then be asked to lay on your back, on a hospital bed or exam table. Electrodes will be placed along your chest, the same way they are placed for an electrocardiogram (ECG--a test to measure the electrical activity of the heart). You will be asked to rest for 15 minutes, and then your heart rhythm will be recorded for 5 minutes. After this first recording, you will begin the relaxation program by listening to an audio recording for about 15 minutes, using headphones. After the relaxation program has ended, your heart rhythm will be recorded for another 5-minute period while you are resting.

You will then be asked to complete the same questionnaire as before.

The entire procedure will take about 45-60 minutes. After this second questionnaire, your participation on this study will be over.

This is an investigational study. Up to 20 people will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Normal cognition (per treating physician's assessment)

Exclusion Criteria:

1. Dementia
2. Psychosis
3. Delirium
4. Not fluent in English
5. Cardiac dysrhythmia
6. Inability to lay supine
7. Pacemaker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Guo, MD, Principal Investigator — U.T. M.D. Anderson Cancer Center Professor
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: U.T. M.D. Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 7/09/2008 through 7/10/2008. All participants recruited at University of Texas MD Anderson Cancer Center.
Pre-assignment Details: One of twenty enrolled participants did not meet eligibility criteria and was excluded from the study.
Period: Overall Study
Arm/Group | Guided Relaxation
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Guided Relaxation
Number analyzed (Participants) | 19
Age Continuous [Median (Full Range); unit: Years] | 57 [25 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Differences Between Pre/Post ESAS Score
Description: Total symptom burden as measured by Edmonton Symptom Assessment Scale (ESAS) in which there are eight visual analog scales (VAS) of 0 to 10, with 10 being most severe. The differences from ESAS baseline (before) to post (after) a 15 minute, one-time, guided relaxation program for each participant assessed, with the average difference in ESAS scores for all participants reported.
Time Frame: Baseline and following completion of HRV recordings and relaxation program (45 - 60 minutes elapsed time)
Population: Analysis included all study participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Guided Relaxation: Heart rate variability (HRV) high frequency (HF) spectral analysis, before and after a 15 minute, one-time, guided relaxation program and summed ESAS scores
Arm/Group | Guided Relaxation
Number analyzed (Participants) | 19
units on a scale | -9.1 (2.4)

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Guided Relaxation
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No